CLINICAL TRIAL: NCT01773174
Title: Single Dose Open-label PK/PD, Safety and Tolerability Study of Dabigatran Etexilate Mesilate Given at the End of Standard Anticoagulant Therapy in Children Aged 1 Year to Less Than 2 Years in Conjunction With Study 1160.89
Brief Title: Pharmacokinetics, Safety and Tolerability of Dabigatran Etexilate Solution in Children 1 to < 2 Years of Age
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.145
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

ARMS (1):
- dabigatran etexilate (Experimental): single dose treatment with dabigatran oral solution
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — age & weight adjusted equivalent of adult dose

SUMMARY:
Study will assess PK/PD parameters and safety and tolerability of the study medication in this age group

ELIGIBILITY:
Inclusion criteria:

1. males or females 1 to less than 2 years of age
2. objective diagnosis of primary venous thromboembolism
3. completion of planned treatment course with low molecular weight heparin or oral anticoagulant for primary venous thromboembolism
4. written informed consent by parent (legal guardian) and patient assent (if applicable)

Exclusion criteria:

1. weight less than 9 kg
2. conditions associated with increased risk of bleeding
3. patients who have any condition that would not allow safe participation in study Note: Further exclusion criteria apply

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Ecarin clotting time (ECT) | one day
Factor IIa inhibition | one day
Incidence of all bleeding events | 30 days
Incidence of all adverse events | 30 days
Plasma concentrations of total dabigatran | one day
Plasma concentrations of free dabigatran | one day
Plasma concentrations of BIBR 1048 BS (Base) | one day
Plasma concentrations of BIBR 951 BS | one day
Plasma concentrations of BIBR 1087 SE (Acid) | one day
Activated prothrombin time (aPTT) | one day

SECONDARY OUTCOMES:
Global assessment of tolerability will be summarized across all patients in the treated set | 30 days
Patient assessment of taste will be summarized across all patients in the treated set | one day
Changes in laboratory and clinical parameters | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (8):
- United States (8):
  - 1160.145.00010 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1160.145.00009 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1160.145.00008 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1160.145.00012 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1160.145.00007 Boehringer Ingelheim Investigational Site, Newark, New Jersey
  - 1160.145.0006 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1160.145.00001 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1160.145.00011 Boehringer Ingelheim Investigational Site, Spokane, Washington